CLINICAL TRIAL: NCT02465450
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of JBT-101 in Cystic Fibrosis
Brief Title: Safety, Tolerability, Pharmacokinetics, and Efficacy of JBT-101 (Lenabasum) in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corbus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: JBT101-CF-001
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
Keywords: JBT-101, Lenabasum, Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lenabasum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- JBT101 (lenabasum) 1 mg (Experimental): JBT-101 1 mg once a day on Days 1-28
  Interventions: Drug: JBT-101 (lenabasum)
- JBT-101 (lenabasum) 5 mg (Experimental): JBT-101 5 mg once a day on Days 1-28
  Interventions: Drug: JBT-101 (lenabasum)
- Placebo (Placebo Comparator): Placebo once a day on Days 1-28.
  Interventions: Other: Placebo
- JBT-101 (lenabasum) 20 mg QD (Experimental): JBT-101 20 mg once a day on Days 29-84.
  Interventions: Drug: JBT-101 (lenabasum)
- JBT-101 (lenabasum) 20 mg BID (Experimental): JBT-101 20 mg twice daily on Days 29-84.
  Interventions: Drug: JBT-101 (lenabasum)
- Placebo BID (Placebo Comparator): Placebo twice daily on Days 29-84.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JBT-101 (lenabasum) — Subjects will receive JBT-101 1 mg qd or JBT-101 5 mg qd on Days 1-28. Subjects will receive either JBT-101 20 mg q am (with placebo q pm) or JBT-101 20 mg twice a day on Days 29-84.
  Arms: JBT-101 (lenabasum) 20 mg BID; JBT-101 (lenabasum) 20 mg QD; JBT-101 (lenabasum) 5 mg; JBT101 (lenabasum) 1 mg
Other: Placebo — Subjects will receive placebo once a day on Days 1-28, placebo q pm on Days 29-84 (with JBT-101 20 mg q am), or placebo bid on Days 29-84.
  Arms: Placebo; Placebo BID

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and efficacy of JBT-101 in adult subjects with cystic fibrosis (CF).

DETAILED DESCRIPTION:
An interventional, double-blind, randomized, placebo-control design will be used to test safety, tolerability, pharmacokinetics, and efficacy of JBT-101 in 70 subjects ≥ 18 and < 65 years of age with documented cystic fibrosis. There will up a screening period of up to 28 days, 84 days treatment period, and 28 days follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of a CF diagnosis as evidenced by 1 or more clinical features consistent with the CF phenotype and 1 or more of the following criteria:

  1. Sweat chloride equal to or greater than 60 mEq/L by quantitative pilocarpine iontophoresis test;
  2. Two well-characterized mutations in the CFTR gene
* FEV1 ≥ 40% predicted corrected
* Stable treatment of CF for 14 days before Visit 1

Exclusion Criteria:

* Severe or unstable CF, such as:

  1. Intravenous antibiotic treatment within 14 days before Visit 1
  2. Treatment with any corticosteroids > 10 mg per day or > 20 mg every other day oral prednisone or equivalent within 14 days before Visit 1
* Any one of the following values for laboratory tests at Screening:

  1. A positive pregnancy test (or at Visit 1);
  2. Hemoglobin < 10 g/dL
  3. Neutrophils < 1.0 x 10~9/L
  4. Platelets < 75 x 10~9/L
  5. Creatinine clearance < 50 ml/min according to modified Cockcroft-Gault equation
  6. Serum transaminases > 2.5 x upper normal limit
  7. Total bilirubin ≥ 1.5 x upper limit of normal
* Any other condition that, in the opinion of the Principal Investigator, is clinically significant and may put the subject at greater safety risk, influence response to study product, or interfere with study assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Chmiel, M.D., Principal Investigator — University Hospitals Cleveland Medical Center, Cleveland, OH; J S Elborn, M.D., Principal Investigator — Queens University, Belfast, Northern Ireland, United Kingdom
Locations (27):
- United States (12):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Long Beach Memorial Medical Center/Miller Children's and Women's Hospital, Long Beach, California
  - National Jewish Health, Denver, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rutgers Robert-Wood Johnson Medical School, New Brunswick, New Jersey
  - North Shore LIJ Health System, New Hyde Park, New York
  - New York Medical College, Valhalla, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital Clinical Care Center, Houston, Texas
- Hôpital Erasme, Brussels, Belgium
- France (3):
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Institution Hôpital Pasteur, Nice
  - Centre de Perharidy, Roscoff
- Germany (2):
  - Christiane Herzog CF-Zentrum Frankfurt am Main, Frankfurt am Main, Hesse
  - UNI Essen Abt.Pneumologie, Essen, North Rhine-Westphalia
- Italy (3):
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - AOUI di Verona - Ospedale Borgo Trento UOC Fibrosi Cistica, Verona
- Poland (4):
  - Szpital Dziecięcy Polanki im. Macieja Płażyńskiego w Gdańsku Spółka z o.o. Poradnia Leczenia Mukowiscydozy, Gdansk
  - Sanatorium Cassia-Villa Medica s.c, Rabka-Zdrój
  - Podkarpacki Ośrodek Pulmunologii i Alergologii, Rzeszów
  - Instytut Gruźlicy i Chorób Płuc I Klinika Chorób Płuc, Warsaw
- United Kingdom (2):
  - Belfast City Hospital, Belfast
  - Queen Elizabeth University Hospital, Glasgow

REFERENCES:
- [Derived] Chmiel JF, Flume P, Downey DG, Dozor AJ, Colombo C, Mazurek H, Sapiejka E, Rachel M, Constantine S, Conley B, Dgetluck N, Dinh Q, White B, Elborn JS; Lenabasum JBT101-CF-001 Study Group. Safety and efficacy of lenabasum in a phase 2 randomized, placebo-controlled trial in adults with cystic fibrosis. J Cyst Fibros. 2021 Jan;20(1):78-85. doi: 10.1016/j.jcf.2020.09.008. Epub 2020 Oct 1. PMID 33011099

RESULTS

PARTICIPANT FLOW:
Groups:
- JBT101 1 mg QD: JBT-101: 1 mg once a day on Days 1-28
- JBT-101 5 mg QD: JBT-101: 5 mg once a day on Days 1-28.
- Placebo QD: Placebo: Subjects received placebo on Days 1 - 28.
- JBT-101 20 mg QD: JBT-101: 20 mg once a day on Days 29 - 84.
  JBT-101: Subjects in this analysis group could have received 1 mg, 5 mg, or placebo during Days 1 - 28.
- JBT-101 20 mg BID: JBT-101: 20 mg twice a day on Days 29 - 84.
  JBT-101: Subjects in this analysis group could have received 1 mg, 5 mg, or placebo during Days 1 - 28.
- Placebo BID: Placebo administered twice daily.
  Subjects in this analysis group received placebo on Days 1 - 28.
Period: Treatment Period 1
Arm/Group | JBT101 1 mg QD | JBT-101 5 mg QD | Placebo QD | JBT-101 20 mg QD | JBT-101 20 mg BID | Placebo BID
Started | 26 | 24 | 35 | 0 | 0 | 0
Completed | 24 | 23 | 34 | 0 | 0 | 0
Not Completed | 2 | 1 | 1 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | JBT101 1 mg QD | JBT-101 5 mg QD | Placebo QD | JBT-101 20 mg QD | JBT-101 20 mg BID | Placebo BID
Started | 0 | 0 | 0 | 30 | 28 | 23
Completed | 0 | 0 | 0 | 27 | 24 | 23
Not Completed | 0 | 0 | 0 | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- JBT101 1 mg QD, 20 mg QD, or 20 mg BID: JBT-101: 1 mg once a day on Days 1-28 and either 20 mg QD or 20 mg BID on Days 29-84.
- JBT-101 5 mg QD,20 mg QD, or 20 mg BID: JBT-101: 5 mg once a day on Days 1-28 and either 20 mg QD or 20 mg BID on Days 29-84.
- Placebo QD,20 mg QD, 20 mg BID, or Placebo BID: Placebo: Subjects received placebo on Days 1 - 28 and either 20 mg QD, 20 mg BID, or Placebo on Days 29-84.
- Total: Total of all reporting groups
Arm/Group | JBT101 1 mg QD, 20 mg QD, or 20 mg BID | JBT-101 5 mg QD,20 mg QD, or 20 mg BID | Placebo QD,20 mg QD, 20 mg BID, or Placebo BID | Total
Number analyzed (Participants) | 26 | 24 | 35 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 2 | 3
  Between 18 and 65 years | 26 | 23 | 33 | 82
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (7.66) | 28.8 (10.40) | 29.2 (8.55) | 28.4 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 18 | 39
  Male | 17 | 12 | 17 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 26 | 22 | 35 | 83
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 25 | 24 | 33 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 171.30 (9.724) | 167.75 (9.192) | 167.82 (8.866) | 168.86 (9.259)
Weight [Mean (Standard Deviation); unit: kg] | 66.98 (14.648) | 64.71 (11.032) | 63.81 (11.806) | 65.03 (12.467)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.735 (3.8582) | 22.976 (3.4182) | 22.608 (3.4672) | 22.751 (3.5381)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events.
Time Frame: 84 days of treatment
Population: These adverse events are based on subjects who entered Treatment Period 2 (n=81). The tabulation of adverse events includes all TEAEs.
Measure: Count of Participants; unit: Participants
Arm/Group | JBT101 1 mg QD | JBT-101 5 mg QD | Placebo QD | JBT-101 20 mg QD | JBT-101 20 mg BID | Placebo BID
Number analyzed (Participants) | 26 | 24 | 35 | 30 | 28 | 23
Participants | 14 | 13 | 15 | 21 | 19 | 14

2. Secondary Outcome: JBT-101 (Lenabasum) Plasma Concentrations on Day 84
Description: Plasma concentrations were reported for the lenabasum 20 mg QD, 20 mg BID, and placebo groups only, at Day 84.
Time Frame: Day 84
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Lenabasum 1 mg QD: Lenabasum: 1 mg once a day on Days 1-28
- Lenabasum 5 mg QD: Lenabasum: 5 mg once a day on Days 1-28.
- Lenabasum 20 mg QD: Lenabasum: 20 mg once a day on Days 29 - 84.
  Lenabasum: Subjects in this analysis group could have received 1 mg, 5 mg, or placebo during Days 1 - 28.
- Lenabasum 20 mg BID: Lenabasum: 20 mg twice a day on Days 29 - 84.
  Lenabasum: Subjects in this analysis group could have received 1 mg, 5 mg, or placebo during Days 1 - 28.
Arm/Group | Lenabasum 1 mg QD | Lenabasum 5 mg QD | Placebo QD | Lenabasum 20 mg QD | Lenabasum 20 mg BID | Placebo BID
Number analyzed (Participants) | 0 | 0 | 0 | 27 | 24 | 23
ng/mL |  |  |  | 249.77 (339.938) | 360.80 (352.772) | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: For treatment groups lenabasum 1 mg QD, lenabasum 5 mg QD and placebo QD, adverse events were collected from Days 1 - 28. For treatment groups lenabasum 20 mg QD, lenabasum 20 mg BID and placebo BID, adverse events were collected from Days 29 - 84.
Arm/Group | JBT101 1 mg QD | JBT-101 5 mg QD | Placebo QD | JBT-101 20 mg QD | JBT-101 20 mg BID | Placebo BID
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/35 | 0/30 | 0/28 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/26 | 2/37 | 3/30 | 2/28 | 1/23
Other Adverse Events (participants affected / at risk) | 13/26 | 13/24 | 15/35 | 21/30 | 19/28 | 14/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JBT101 1 mg QD (N=26) | JBT-101 5 mg QD (N=26) | Placebo QD (N=37) | JBT-101 20 mg QD (N=30) | JBT-101 20 mg BID (N=28) | Placebo BID (N=23)
hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Thrombosis in device (General disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JBT101 1 mg QD (N=26) | JBT-101 5 mg QD (N=24) | Placebo QD (N=35) | JBT-101 20 mg QD (N=30) | JBT-101 20 mg BID (N=28) | Placebo BID (N=23)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 6 (7) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Cognitive disorder (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 4 (5) | 1 (1) | 3 (4) | 4 (4)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 | 1 (2) | 0
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 (2) | 0 | 0
Lethargy (Nervous system disorders) | 1 (1) | 0 | 0 (0) | 2 (2) | 1 (1) | 0
Haemoptysia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (6) | 3 (3) | 0
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Gastroeosophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 | 1 (1) | 0
Sweat discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Gastrostomy (Surgical and medical procedures) | 0 | 0 | 1 (1) | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1)
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 (2) | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Bradykinesia (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Stupor (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Thrombosis (General disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Chest discomfort (General disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other